CLINICAL TRIAL: NCT05015998
Title: A Non-interventional Evaluation of the ePidemiology of anEmia Associated With chroNic Kidney Disease in Patients in Primary Care Using The Stockholm CREAtinine Measurement (SCREAM) Register
Brief Title: A Study to Evaluate the ePidemiology of anEmia Associated With chroNic Kidney Disease in Patients in Primary Care Using The Stockholm CREAtinine Measurement (SCREAM) Register
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 1517-MA-1569
Record Dates: First submitted 2021-08-15; First posted 2021-08-23 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; SCREAM database
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-dialysis dependent patients with CKD stage 3-5: A cohort of patients will be created from the Stockholm CREAtinine Measurement (SCREAM) cohort based on the eligibility criteria.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Epidemiology of anemia associated with chronic kidney disease, rather than to evaluate specific drugs

SUMMARY:
The objectives of this analysis is to determine the incidence of anemia occurring in patients with chronic kidney disease (CKD) in primary care (i.e. prior to any eventual referral to nephrology care). This analysis also evaluates patient characteristics, anemia treatment and associated cardiovascular risk.

DETAILED DESCRIPTION:
Data will be derived from the Stockholm CREATinine Measurement (SCREAM) cohort, a repository of laboratory data of individuals residing and accessing healthcare in the region of Stockholm and who underwent a creatinine assessment between 2012 - 2018.

ELIGIBILITY:
Inclusion Criteria:

* Patient entered in SCREAM between 2012 and 2018
* With two consecutive plasma-creatinine test(s) indicating an estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m^2
* With at least one eligible Hb after eGFR < 60 mL/min/1.73 m^2. The date of the first eligible Hb test is the study entry point/index date of the study.

Exclusion Criteria:

* Patient who has had a recent pregnancy or childbirth (issued diagnosis within 2 years prior to index date).
* Patient with ongoing/recent cancer (diagnosed within the previous 3 years), haematological diseases or leukaemia.
* Patient with chronic infections (hepatitis, tuberculosis, or human immunodeficiency virus [HIV]); note by definition chronic infections are chronic and look back period will be to 1997.
* Patients with anemia at baseline (index date), defined by an anemia diagnosis in the year prior, a baseline Hb value within the anemia range according to the WHO definition, or the presence of a recent dispensation of ESA or iron (up to six months prior).
* Patient referred to nephrologist within the previous 2 years from cohort entry/ index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary data source will be the Stockholm CREAtinine Measurement (SCREAM) cohort. This is a cohort comprising Swedish citizens residing in or accessing healthcare in Stockholm county with a valid personal identification number and a creatinine measurement taken between 2006 - 2018. Records of patients meeting inclusion criteria, in this healthcare utilization cohort will be linked to national Swedish registries including the Regional healthcare utilization registry, the national Patient Registry and the National Prescribed Drugs Registry.
Sampling Method: Non-Probability Sample
Enrollment: 45637 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence rate of anemia in adults with non-dialysis dependent CKD stage 3-5 in primary care | 6 years at maximum
  Anemia will be defined as the composite of: a diagnosis of anemia, a haemoglobin (Hb) measurement within the defined range for anemia followed by iron (oral or intravenous [IV]) or erythropoietin-simulating agent (ESA) treatment within 3 months, a Hb measurement within the defined range for anemia followed by another low Hb measurement >3 months apart. Anemia as an outcome will be defined by current World Health Organization (WHO) definitions (Hb < 12 g/dL or 7.45 mmol/L for female and < 13 g/dL or 8.07 mmol/L for male). The incidence rate of anemia will be calculated as the number of new cases divided by person-time of CKD stage 3-5 patients who were "at risk" of becoming an incident anemia case.

SECONDARY OUTCOMES:
Baseline characteristics associated with anemia occurrence in unreferred CKD stage 3-5 patients | On Day 1
  The prevalence of different baseline characteristics of interest will be summarized.
Comorbidities associated with anemia occurrence in unreferred CKD stage 3-5 patients | On Day 1
  The prevalence of different comorbidities of interest will be summarized.
Proportion of patients who initiated anemia treatment after incident of anemia | 6 months
  Anemia treatment initiated within 6 months after development of anemia can include oral iron, IV iron, or erythropoietin-simulating agent (ESA).
Correlation of incident anemia and the risk of major adverse cardiac events (MACE) events in patients in anemia exposed period | 7 years at maximum
  MACE will be defined as all-cause mortality, non-fatal stroke and non-fatal myocardial infarction. Anemia exposed period is from incident anemia until event or end of follow-up.
Correlation of incident anemia and the risk of major adverse cardiac events (MACE) events in patients in anemia non-exposed period | 7 years at maximum
  MACE will be defined as all-cause mortality, non-fatal stroke and non-fatal myocardial infarction. The non-exposed period is from baseline (no anemia) until event or the time of anemia development.
Correlation of incident anemia and the risk of MACE+ in patients in anemia exposed period | 7 years at maximum
  MACE+ will be defined as any record defining MACE, plus hospitalization for unstable angina or hospitalization for congestive heart failure. Anemia exposed period is from incident anemia until event or end of follow-up.
Correlation of incident anemia and the risk of MACE+ in patients in non-anemia exposed period | 7 years at maximum
  MACE+ will be defined as any record defining MACE, plus hospitalization for unstable angina or hospitalization for congestive heart failure. The non-exposed period is from baseline (no anemia) until event or the time of anemia development.
Correlation of incident anemia and the risk of death in patients with anemia | 7 years at maximum
  Proportion of death in patients with anemia

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe Ltd.
Locations (1):
- SE46001, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://www.clinicaltrials.astellas.com/study/1517-MA-1569/